CLINICAL TRIAL: NCT06606392
Title: Effect of Biodex Balance Training and Short Foot Exercise on Myoelectric Activity of Paraspinal Muscles in Subjects with Flexible Flatfoot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: MTI University (Other)
Responsible Party: Principal Investigator, Hager Mahmoud mohamed elsayed, Assistant lecturer basic science department of faculty of physical therapy modern university for technology and science, MTI University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BSM
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Flat Foot
Keywords: Flat foot, Myoelectric activity, Biodex balance
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Other): Group A 30 subjects will receive short foot exercise and stretching exercise gastrocnemius, soleus muscle and planter fascia stretch.
  Interventions: Other: Short Foot Exercise
- Group B (Experimental): Group B will receive Biodex balance training and short foot exercise.
  Interventions: Device: Biodex balance system; Other: Short Foot Exercise

INTERVENTIONS:
Device: Biodex balance system — The Biodex Balance System has a wide range of clinical applications and provides objective measures from testing that can be used to establish progressions and discharge criteria, as well as be part of a comprehensive Fall Risk Assessment or Fall Screening Program. Balance ability can be assessed either statically or dynamically, as well as bilaterally and unilaterally. It also allows for bilateral comparisons between involved and uninvolved limbs.
  Arms: Group B
Other: Short Foot Exercise — Short foot exercise is used as a therapeutic exercise to strengthen intrinsic foot muscles and used as training to create an MLA. It helps improve the balance in functional movement of FF subjects, decreases navicular drop (ND) through intrinsic muscle activation, supports navicular stability, and improves balance

SUMMARY:
The goal of this study is to see the effect of the combination of biodex balance system and short foot exercise in the treatment of subjects with flexible flat foot. The main question is the effect of biodex balance training and short foot exercise on myoelectric activity of subjects with flexible flat foot experimental participant will receive biodex balance system exercise and short foot exercise for 4 weeks controlled participant will receive short foot exercise and stretching exercise for 4 weeks Assessment will be done pre and post treatment by using Navicular drop test Myoelectric activity of paraspinal muscle Dynamic balance Pain severity Functional ankle instability inder

ELIGIBILITY:
Inclusion Criteria:

* 1) Sixty subjects from both gender with bilateral flexible flat foot will be selected with their age between 18 to 30Years old 2) Body Mass Index (BMI) was ranging from 18 to 25 kg/m2 3) The participants were eligible to be included if had bilaterally FFF according to the navicular drop test 4) Required participant to have been diagnosed (by an orthopedist) with flexible flat foot

Exclusion Criteria:

* Repeated lower extremity injuries as fractures or deformities. 2) History of surgery to the lower extremity. 3) History of cerebral concussions, and visual or vestibular disorders. 4) Any neurological deficit affecting balance. 5) Any medication can affect the balance 6) Any problem of lumbar spine( disc,spondylolisthrsis)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Muscle myoelectric activity | 4 weeks
  myoelectric activity of paraspinal muscles measured by surface electromygraphy
Foot print pressure | 4 weeks
  Using myopressure force platform to measure average peak planter pressure
Dynamic balance | 4 weeks
  Biodex balance system will be used to assess balance before and after treatment
Functional ankle instability index | 4 weeks
  Cumberland Ankle Instability Tool The CAIT is a nine-item questionnaire intended to identify and grade ankle instability
Pain severity | 4 weeks
  Evaluation of lower back pain severity by using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Ragia M kamal, Doctoral, Principal Investigator — professor of physical therapy , cairo university; Naglaa F Awes, Doctoral, Principal Investigator — Assistant professor of physical therapy cairo universiy; Hend H Mohamed, Doctoral, Principal Investigator — Lecturer of physical therapy cairo university; Hager M Elsayed, Master, Principal Investigator — assistant lecturer of faculty of physical therapy, modern university for technology and science
Locations (1):
- Modern university for technology and science, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Aenumulapalli A, Kulkarni MM, Gandotra AR. Prevalence of Flexible Flat Foot in Adults: A Cross-sectional Study. J Clin Diagn Res. 2017 Jun;11(6):AC17-AC20. doi: 10.7860/JCDR/2017/26566.10059. Epub 2017 Jun 1. PMID 28764143